CLINICAL TRIAL: NCT04594460
Title: A Clinical Trial to Evaluate the Efficacy and Safety of Hydrogen-oxygen Mixed Gas Inhalation in Convalescent Severe/Critically Ill Patients With Novel Coronavirus Pneumonia (COVID-19)
Brief Title: Hydrogen-oxygen Gas Mixture Inhalation in Patients With Convalescent Coronavirus Disease 2019 (COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, Doctor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMS-H-03-101
Record Dates: First submitted 2020-10-19; First posted 2020-10-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Hydrogen-oxygen Gas; AMS-H-03
Keywords: Covid19; Hydrogen-oxygen Gas; AMS-H-03
MeSH Terms: conditions — COVID-19 | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: Subjects in the experimental arm and the control arm will receive hydrogen-oxygen mixed gas inhalation (Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03, output: 3 L/min (hydrogen concentration: 66.7%, oxygen concentration: 33.3%)) and oxygen inhalation (OLO-1 Medical Molecular Sieve Oxygen Generator, output: 3 L/min (oxygen concentration: 33.3%), Shanghai Ouliang Medical Devices Co., Ltd.), respectively; the targeted treatment duration will be 8 hours per day, for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is conducted in a double-blind design with a primary unblinding, and a terminal unblinding is performed after data review, database lock, and finalization of the statistical analysis plan.
  Both the investigational device (AMS-H-03 Hydrogen-Oxygen Generator with Nebulizer) and the control device (OLO-1 Medical Molecular Sieve Oxygen Generator) were placed in the shell with the same appearance, with the same operating interface and only ventilation function. During the treatment, neither the investigator nor the subject would be aware of the treatment allocation The study devices will be masked by independent non-blinded personnel of the statistical company according to the corresponding operating procedures, and no specific personnel participating in the clinical operation shall be present during the process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental Group (Experimental): the experimental arm will receive hydrogen-oxygen mixed gas inhalation (Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03, output: 3 L/min (hydrogen concentration: 66.7%, oxygen concentration: 33.3%)) ,the treatment duration will be 8 hours per day, for 12 weeks.
  Interventions: Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03
- Control Group (Active Comparator): the control arm will receive oxygen inhalation (OLO-1 Medical Molecular Sieve Oxygen Generator, output: 3 L/min (oxygen concentration: 33.3%), Shanghai Ouliang Medical Devices Co., Ltd.)the treatment duration will be 8 hours per day, for 12 weeks.
  Interventions: Device: OLO-1 Medical Molecular Sieve Oxygen Generator

INTERVENTIONS:
Device: Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03 — the experimental arm will receive hydrogen-oxygen mixed gas inhalation (Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03, output: 3 L/min (hydrogen concentration: 66.7%, oxygen concentration: 33.3%)) ,the treatment duration will be 8 hours per day, for 12 weeks.
  Arms: experimental Group
Device: OLO-1 Medical Molecular Sieve Oxygen Generator — the control arm will receive oxygen inhalation (OLO-1 Medical Molecular Sieve Oxygen Generator, output: 3 L/min (oxygen concentration: 33.3%), Shanghai Ouliang Medical Devices Co., Ltd.)the treatment duration will be 8 hours per day, for 12 weeks.
  Arms: Control Group

SUMMARY:
This study is a multicenter, randomized, open, parallel-controlled study. Qualified subjects will randomly be assigned to the experimental arm or the control arm according to the ratio of 1:1, with age (> 60 years or ≤ 60 years), smoking status (yes/no) and forced expiratory volume in one second/prediction (FEV1 %pred > 60% or ≤ 60%) as the random stratification factors.

DETAILED DESCRIPTION:
Subjects in the experimental arm and the control arm will receive hydrogen-oxygen mixed gas inhalation (Hydrogen-Oxygen Generator with Nebulizer, AMS-H-03, output: 3 L/min (hydrogen concentration: 66.7%, oxygen concentration: 33.3%)) and oxygen inhalation (OLO-1 Medical Molecular Sieve Oxygen Generator, output: 3 L/min (oxygen concentration: 33.3%), Shanghai Ouliang Medical Devices Co., Ltd.), respectively; the treatment duration will not be less than 8 hours per day, for 12 weeks.

Subjects in the experimental arm and the control arm will also receive other medications (excluding antiviral drugs) by the investigator as clinically indicated. Six visits are required for each subject in this study, including Visit 1 (D-7~-1), Visit 2 (D1), Visit 3 (D14±3d), Visit 4 (D28±3d), Visit 5 (D56±7d), Visit 6 (D84±7d).

ELIGIBILITY:
Inclusion Criteria:

* 1） Male or female, aged between 18 and 75 (including boundary values) at screening.

  2) Severe or critically ill patients who have been diagnosed with a novel coronavirus during hospitalization (COVID-19).

  3) After treatment, the patients have met the discharge criteria of "COVID-19 Diagnosis and Treatment Guideline", and the time from hospital discharge is at least 1 month at the time of enrollment. The clinical symptoms of the subjects did not worsen significantly as compared with that at the time of discharge, and the COVID-19 nucleic acid test results are negative for at least 2 consecutive times (one of which could be the nucleic acid test before discharge).

  4) Forced vital capacity/per predicted (FVC% pred) ≥ 50%. 5) 50% ≤ FEV1 %pred ≤80%。 6) Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures. Understands and agrees to comply with planned study procedures.

  7) Agrees not to participate in other drug/device studies until the study is completed.

Exclusion Criteria:

* 1) With one of the following respiratory diseases:

  1. Subjects with asthma history, or cannot rule out asthma based on the diagnosis of investigator;
  2. Subjects with chronic obstructive pulmonary disease (COPD);
  3. Subjects with following respiratory diseases such as active tuberculosis, lung cancer, sarcoidosis, pulmonary hypertension, pneumothorax, uncontrolled pleural effusion through intervention, pulmonary embolism, etc.;
  4. Lung volume reduction: subjects have had lung volume reduction surgery, pulmonary lobectomy, or bronchoscopic lung volume reduction surgery.

     2) Subjects with pulmonary heart disease. 3) Patients who are scheduled for elective surgery during the study period, such as thoracic and abdominal major surgery.

     4) Subjects, judged by investigators, with previous or current diseases, which may affect the participation in this study or the outcome of this study: such as cancer, diseases of heart, liver, kidney, hematopoietic system and other vital organs or systems, etc.

     5) Patients who have undergone surgery within 1 month prior to screening and have not fully recovered.

     6) Occurrence of congestive heart failure, uncontrolled or unstable angina or myocardial infarction, cerebrovascular accident, or history of pulmonary embolism within 6 months prior to screening.

     7) Patients with active tuberculosis infection within 12 months prior to screening.

     8) Pregnancy or lactating women, or women of childbearing potential not agree to either abstinence or use at least one primary form of contraception from the time of screening till the study is completed.

     9) Subjects with mental disorders or other conditions that are unable to cooperate effectively with the conduct of the clinical trial.

     10) Subjects intolerance to inhalation therapy. 11) Others whom the investigator or sub-investigator judged inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
(VO2max) | The change from baseline in maximum oxygen consumption (VO2max) at maximum exercise load at Week 12 of treatment.
  The change from baseline in maximum oxygen consumption (VO2max) at maximum exercise load at Week 12 of treatment.

SECONDARY OUTCOMES:
(VO2max) | The change from baseline in maximum oxygen consumption (VO2max) at maximum exercise load at Week 4 of treatment.
  The change from baseline in maximum oxygen consumption (VO2max) at maximum exercise load at Week 4 of treatment.
(VO2max) | The change from baseline in maximum oxygen consumption (VO2max) at maximum exercise load at Week 8 of treatment.
  The change from baseline in maximum oxygen consumption (VO2max) at maximum exercise load at Week 8 of treatment.
(VE /VCO2) | Differences in the change from baseline in ventilatory equivalent for carbon dioxide (VE /VCO2) at maximum exercise load at Week 4 of treatment.
  Differences in the change from baseline in ventilatory equivalent for carbon dioxide (VE /VCO2) at maximum exercise load at Week 4 of treatment.
(VE /VCO2) | Differences in the change from baseline in ventilatory equivalent for carbon dioxide (VE /VCO2) at maximum exercise load at Week 8 of treatment.
  Differences in the change from baseline in ventilatory equivalent for carbon dioxide (VE /VCO2) at maximum exercise load at Week 8 of treatment.
(VE /VCO2) | Differences in the change from baseline in ventilatory equivalent for carbon dioxide (VE /VCO2) at maximum exercise load at Week 12 of treatment.
  Differences in the change from baseline in ventilatory equivalent for carbon dioxide (VE /VCO2) at maximum exercise load at Week 12 of treatment.
(VE /VO2) | Differences in the change from baseline in ventilatory equivalent for oxygen (VE /VO2) at maximum exercise load at Week 4 of treatment.
  Differences in the change from baseline in ventilatory equivalent for oxygen (VE /VO2) at maximum exercise load at Week 4 of treatment.
(VE /VO2) | Differences in the change from baseline in ventilatory equivalent for oxygen (VE /VO2) at maximum exercise load at Week 8 of treatment.
  Differences in the change from baseline in ventilatory equivalent for oxygen (VE /VO2) at maximum exercise load at Week 8 of treatment.
(VE /VO2) | Differences in the change from baseline in ventilatory equivalent for oxygen (VE /VO2) at maximum exercise load at Week 12 of treatment.
  Differences in the change from baseline in ventilatory equivalent for oxygen (VE /VO2) at maximum exercise load at Week 12 of treatment.
(VO2 /HR) | Differences in the change from baseline in oxygen pulse (VO2 /HR) at maximum exercise load at Week 4 of treatment.
  Differences in the change from baseline in oxygen pulse (VO2 /HR) at maximum exercise load at Week 4 treatment.
(VO2 /HR) | Differences in the change from baseline in oxygen pulse (VO2 /HR) at maximum exercise load at Week 8 of treatment.
  Differences in the change from baseline in oxygen pulse (VO2 /HR) at maximum exercise load at Week 8 of treatment.
(VO2 /HR) | Differences in the change from baseline in oxygen pulse (VO2 /HR) at maximum exercise load at Week 12 of treatment.
  Differences in the change from baseline in oxygen pulse (VO2 /HR) at maximum exercise load at Week 12 of treatment.
(P (A-a) O2) | The change from baseline in the alveolar-arterial oxygen tension gradient (P (A-a) O2) at maximum exercise load at Week 4 of treatment.
  The change from baseline in the alveolar-arterial oxygen tension gradient (P (A-a) O2) at maximum exercise load at Week 4 of treatment.
(P (A-a) O2) | The change from baseline in the alveolar-arterial oxygen tension gradient (P (A-a) O2) at maximum exercise load at Week 8 of treatment.
  The change from baseline in the alveolar-arterial oxygen tension gradient (P (A-a) O2) at maximum exercise load at Week 8 of treatment.
(P (A-a) O2) | The change from baseline in the alveolar-arterial oxygen tension gradient (P (A-a) O2) at maximum exercise load at Week 12 of treatment.
  The change from baseline in the alveolar-arterial oxygen tension gradient (P (A-a) O2) at maximum exercise load at Week 12 of treatment.
(P (a-et) CO2) | The change from baseline in the arterial-to-end-tidal CO2 difference (P (a-et) CO2) at maximum exercise load at Week 4 of treatment.
  The change from baseline in the arterial-to-end-tidal CO2 difference (P (a-et) CO2) at maximum exercise load at Week 4 of treatment.
(P (a-et) CO2) | The change from baseline in the arterial-to-end-tidal CO2 difference (P (a-et) CO2) at maximum exercise load at Week 8 of treatment.
  The change from baseline in the arterial-to-end-tidal CO2 difference (P (a-et) CO2) at maximum exercise load at Week 8 of treatment.
(P (a-et) CO2) | The change from baseline in the arterial-to-end-tidal CO2 difference (P (a-et) CO2) at maximum exercise load at Week 12 of treatment.
  The change from baseline in the arterial-to-end-tidal CO2 difference (P (a-et) CO2) at maximum exercise load at Week 12 of treatment.
maximum exercise power | The change from baseline in maximum exercise power at Week 4 of treatment.
  The change from baseline in maximum exercise power at Week 4 of treatment.
maximum exercise power | The change from baseline in maximum exercise power at Week 8 of treatment.
  The change from baseline in maximum exercise power at Week 8 of treatment.
maximum exercise power | The change from baseline in maximum exercise power at Week 12 of treatment.
  The change from baseline in maximum exercise power at Week 12 of treatment.
RER | The change from baseline in respiratory quotient (RER) at maximum exercise load at Week 4 of treatment.
  The change from baseline in respiratory quotient (RER) at maximum exercise load at Week 4 of treatment.
RER | The change from baseline in respiratory quotient (RER) at maximum exercise load at Week 8 of treatment.
  The change from baseline in respiratory quotient (RER) at maximum exercise load at Week 8 of treatment.
RER | The change from baseline in respiratory quotient (RER) at maximum exercise load at Week 12 of treatment.
  The change from baseline in respiratory quotient (RER) at maximum exercise load at Week 12 of treatment.
The change from baseline in total exercise duration at maximum exercise load at Week 4 of treatment. | The change from baseline in total exercise duration at maximum exercise load at Week 4 of treatment.
  The change from baseline in total exercise duration at maximum exercise load at Week 4 of treatment.
The change from baseline in total exercise duration at maximum exercise load at Week 8 of treatment. | The change from baseline in total exercise duration at maximum exercise load at Week 8 of treatment.
  The change from baseline in total exercise duration at maximum exercise load at Week 8 of treatment.
The change from baseline in total exercise duration at maximum exercise load at Week 12 of treatment. | The change from baseline in total exercise duration at maximum exercise load at Week 12 of treatment.
  The change from baseline in total exercise duration at maximum exercise load at Week 12 of treatment.
(SpO2) | The change from baseline in fingertip oxygen saturation (SpO2) at rest and without oxygen inhalation at Week 4 of treatment.
  The change from baseline in fingertip oxygen saturation (SpO2) at rest and without oxygen inhalation at Week 4 of treatment.
(SpO2) | The change from baseline in fingertip oxygen saturation (SpO2) at rest and without oxygen inhalation at Week 8 of treatment.
  The change from baseline in fingertip oxygen saturation (SpO2) at rest and without oxygen inhalation at Week 8 of treatment.
(SpO2) | The change from baseline in fingertip oxygen saturation (SpO2) at rest and without oxygen inhalation at Week 12 of treatment.
  The change from baseline in fingertip oxygen saturation (SpO2) at rest and without oxygen inhalation at Week 12 of treatment.
(mMRC) | The change from baseline in the modified Medical Research Council (mMRC) Dyspnea Scale score at week 4 of treatment.
  The change from baseline in the modified Medical Research Council (mMRC) Dyspnea Scale score at week 4 of treatment.
(mMRC) | The change from baseline in the modified Medical Research Council (mMRC) Dyspnea Scale score at week 8 of treatment.
  The change from baseline in the modified Medical Research Council (mMRC) Dyspnea Scale score at week 8 of treatment.
(mMRC) | The change from baseline in the modified Medical Research Council (mMRC) Dyspnea Scale score at week 12 of treatment.
  The change from baseline in the modified Medical Research Council (mMRC) Dyspnea Scale score at week 12 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-jie Guan, PhD, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (2):
- China (2):
  - Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kannan S, Shaik Syed Ali P, Sheeza A, Hemalatha K. COVID-19 (Novel Coronavirus 2019) - recent trends. Eur Rev Med Pharmacol Sci. 2020 Feb;24(4):2006-2011. doi: 10.26355/eurrev_202002_20378. PMID 32141569
- [Background] Chinese Clinical Guidance for COVID-19 Penumonia Diagnosis and Treatment (7th edition)
- [Background] Huang X, Wei F, Hu L, Wen L, Chen K. Epidemiology and Clinical Characteristics of COVID-19. Arch Iran Med. 2020 Apr 1;23(4):268-271. doi: 10.34172/aim.2020.09. PMID 32271601
- [Background] Li LQ, Huang T, Wang YQ, Wang ZP, Liang Y, Huang TB, Zhang HY, Sun W, Wang Y. COVID-19 patients' clinical characteristics, discharge rate, and fatality rate of meta-analysis. J Med Virol. 2020 Jun;92(6):577-583. doi: 10.1002/jmv.25757. Epub 2020 Mar 23. PMID 32162702
- [Background] Li K, Wu J, Wu F, Guo D, Chen L, Fang Z, Li C. The Clinical and Chest CT Features Associated With Severe and Critical COVID-19 Pneumonia. Invest Radiol. 2020 Jun;55(6):327-331. doi: 10.1097/RLI.0000000000000672. PMID 32118615
- [Background] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Background] Zhou ZQ, Zhong CH, Su ZQ, Li XY, Chen Y, Chen XB, Tang CL, Zhou LQ, Li SY. Breathing Hydrogen-Oxygen Mixture Decreases Inspiratory Effort in Patients with Tracheal Stenosis. Respiration. 2019;97(1):42-51. doi: 10.1159/000492031. Epub 2018 Sep 18. PMID 30227423
- [Background] Yang Y, Zhu Y, Xi X. Anti-inflammatory and antitumor action of hydrogen via reactive oxygen species. Oncol Lett. 2018 Sep;16(3):2771-2776. doi: 10.3892/ol.2018.9023. Epub 2018 Jun 26. PMID 30127861
- [Background] Zhang N, Deng C, Zhang X, Zhang J, Bai C. Inhalation of hydrogen gas attenuates airway inflammation and oxidative stress in allergic asthmatic mice. Asthma Res Pract. 2018 Mar 15;4:3. doi: 10.1186/s40733-018-0040-y. eCollection 2018. PMID 29568538
- [Background] Guan WJ, Wei CH, Chen AL, Sun XC, Guo GY, Zou X, Shi JD, Lai PZ, Zheng ZG, Zhong NS. Hydrogen/oxygen mixed gas inhalation improves disease severity and dyspnea in patients with Coronavirus disease 2019 in a recent multicenter, open-label clinical trial. J Thorac Dis. 2020 Jun;12(6):3448-3452. doi: 10.21037/jtd-2020-057. No abstract available. PMID 32642277
- [Background] Ong KC, Ng AW, Lee LS, Kaw G, Kwek SK, Leow MK, Earnest A. Pulmonary function and exercise capacity in survivors of severe acute respiratory syndrome. Eur Respir J. 2004 Sep;24(3):436-42. doi: 10.1183/09031936.04.00007104. PMID 15358703